CLINICAL TRIAL: NCT00060749
Title: Investigation of the Effect of Dietary Docosahexaenoic Acid (DHA) Supplementation on Macular Function in Subjects With Autosomal Dominant Stargardt-Like and Autosomal Recessive Stargardt Macular Dystrophy
Brief Title: Effect of DHA Supplements on Macular Function in Patients With Stargardt Macular Dystrophy and Stargardt-like Macular Dystrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030179; 03-EI-0179
Record Dates: First submitted 2003-05-09; First posted 2003-05-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-10

CONDITIONS: Macular Degeneration
Keywords: Stargardt; Macular Dystrophy; ELOVL4; DHA; Stargardt's Disease; Autosomal Dominant Macular Dystrophy; Autosomal Recessive Macular Dystrophy
MeSH Terms: conditions — Macular Degeneration; Erythrokeratodermia with ataxia; Stargardt Disease | interventions — Docosahexaenoic Acids; Dietary Supplements

INTERVENTIONS:
Drug: Docosahexaenoic Acid (DHA) Dietary Supplement

SUMMARY:
This study will evaluate whether docosahexaenoic acid (DHA) dietary supplementation can improve macular function in patients with Stargardt macular dystrophy and Stargardt-like macular dystrophy. Stargardt macular dystrophy is a recessive inherited trait that causes a severe form of macular degeneration. (The macula is the center part of the retina in the back of the eye that is responsible for fine vision.) The disorder begins in late childhood and progresses to a significant decrease in central vision. One of the earliest signs of the disorder is accumulation in and under the macula of a fatty pigment called lipofuscin. Stargardt-like macular dystrophy is a dominant inherited trait involving loss of central vision, but it begins later than Stargardt macular dystrophy, and the accumulation of lipofuscin extends beyond the central region of the macula. DHA is a fatty acid that is essential for normal brain and eye development. It is normally found in the diet, but not in large amounts. Supplements may help prevent or slow the progression of some eye diseases.

Patients with autosomal dominant Stargardt-like macular dystrophy or autosomal recessive Stargardt macular dystrophy are eligible for this study. Candidates will be screened with the following tests and procedures:

* Medical history and physical examination.
* Blood test to measure levels of DHA and vitamins.
* Eye examination: The patient's vision and eye pressure are tested, then the pupils are dilated to examine structures inside the eye. Photographs are also taken.
* Visual field test: The patient looks at a tiny spot of light projected onto a white screen and is asked to note when other lights appear at other places on the screen.
* Electroretinogram (ERG): An electrode (small silver disk) is taped to the patient's forehead. Drops are given to numb the eyes and special contact lenses are inserted in the eyes. For the first part of the test, the patient looks at the center of a black and white checkerboard screen that flickers for 30 seconds at a time. This is repeated 16 or more times. For the second part of the test, the patient looks inside a sphere, in which flashes of light flicker for 20 seconds at a time. This is repeated four or more times. The contact lenses sense small electrical signals generated by the retina during the tests.

Participants will begin taking DHA capsules or a placebo (look-alike capsules with no active ingredient) from 1 week to 3 months after enrolling in the study and will repeat several of the screening tests at follow-up visits scheduled 3, 6, 9, 12, and 15 months after they start taking the capsules. They will also be interviewed about any treatment side effects.

DETAILED DESCRIPTION:
We propose to undertake a double-masked, randomized, placebo-controlled, crossover study on the effect of docosahexaenoic acid (DHA) dietary supplementation in subjects with macular dystrophy to determine whether DHA can improve macular function. Subjects will receive either oral DHA supplementation (5x200 mg BID, 2,000 mg/day) or placebo. Subjects will 'crossover' to the opposite treatment twice during this study. Primary outcomes will measure the change in macular function during periods with and without DHA supplementation.

Zhang and colleagues found a mutation in the gene, ELOVL4 (elongation of the very long chain fatty acid-4), in individuals with Stargardt-like macular dystrophy. The gene is presumed to function in the pathway of synthesis of very long chain polyunsaturated fatty acids, including DHA. DHA is the major very long chain polyunsaturated fatty acid of the retina. As our North American diet is poor in DHA, we hypothesize that a DHA dietary supplement might improve macular function in individuals with the ELOVL4 mutation. Since the effect of DHA supplementation may be non-specific, we propose to study a second cohort with Stargardt macular dystrophy, which has a different genotype involving a different metabolic pathway in the eye, but presents with a similar phenotype. Two cohorts of up to 10 subjects for analysis will be recruited from patients with either Stargardt-like macular dystrophy or Stargardt macular dystrophy.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to enroll in this study, a prospective participant must satisfy the following inclusion criteria.

1. Understand and sign the informed consent.
2. Able to comply with all study procedures (likely to exclude participants less than 10 years of age, but not necessarily).

   Autosomal Recessive Stargardt Macular Dystrophy Participants (must be observed in at least one study eye):
3. Have a pattern of inheritance that indicates autosomal recessive inheritance.
4. Have a phenotype consistent with the diagnosis of autosomal recessive Stargardt macular dystrophy including the following clinical features: fundus examination showing bilateral central maculopathy and/or fundus flecks, or characteristic changes on an intravenous fluorescein angiogram.

   Autosomal Dominant Stargardt-like Macular Dystrophy Participants (must be observed in at least one study eye):
5. Have a pattern of inheritance that indicates autosomal dominant inheritance.
6. Have a phenotype consistent with the diagnosis of Stargardt-like macular dystrophy that may include: fundus examination showing bilateral central maculopathy and fundus flecks confined to the central macula, or intravenous fluorescein angiogram.

EXCLUSION CRITERIA:

To be eligible to enroll in this study, a prospective participant must not satisfy any of the following exclusion criteria.

1. Have a non-recordable multi-focal ERG.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22
Dates: Start 2003-05-05; Study Completion 2007-12-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Zhang K, Kniazeva M, Han M, Li W, Yu Z, Yang Z, Li Y, Metzker ML, Allikmets R, Zack DJ, Kakuk LE, Lagali PS, Wong PW, MacDonald IM, Sieving PA, Figueroa DJ, Austin CP, Gould RJ, Ayyagari R, Petrukhin K. A 5-bp deletion in ELOVL4 is associated with two related forms of autosomal dominant macular dystrophy. Nat Genet. 2001 Jan;27(1):89-93. doi: 10.1038/83817. PMID 11138005